CLINICAL TRIAL: NCT01251354
Title: A Phase II, International, Multicenter, Open-label, Proof of Concept Study of BN83495 in Postmenopausal Women With Advanced, Metastatic or Recurrent Oestrogen Receptor (ER) Positive Endometrial Carcinoma Who Have Received One Line of Chemotherapy in the Adjuvant or Metastatic Setting.
Brief Title: Study of BN83495 in Post-menopausal Women With Endometrial Cancer Post-chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The futility analysis of study NCT00910091 in patients with endometrial cancer shows that the primary endpoint will not be reached.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X-52-58064-007
Record Dates: First submitted 2010-11-23; First posted 2010-12-01 (Estimated); Results first posted 2015-09-02 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — irosustat

ARMS (1):
- BN83495 (Experimental)
  Interventions: Drug: BN83495

INTERVENTIONS:
Drug: BN83495 — 1 tablet of 40 mg, oral, daily until progression or death or unacceptable toxicity develops

SUMMARY:
The purpose of the protocol is to determine the effect of BN83495 on the progression of endometrial cancer with estrogen receptor in post menopausal women who had previously received chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study related procedures.
* postmenopausal or ovariectomised female patient over 18 years of age.
* histologically confirmed diagnosis of ER positive endometrial carcinoma in the primary tumour or metastatic disease
* patient has received one line of chemotherapy prior to enrolment in the adjuvant or in the metastatic setting (including chemoradiotherapy) and progressed after this line of chemotherapy
* patient has at least one measurable disease site (RECIST criteria version 1.1)

Exclusion Criteria:

* patient has received hormone therapy for endometrial cancer in the adjuvant or metastatic setting
* patient has received more than one line of chemotherapy in the adjuvant or metastatic setting
* patient was treated with any other investigational agent within the 3 weeks before study entry.
* patient has ongoing cardiac dysrhythmias grade ≥2, atrial fibrillation of any grade (NCI CTCAE) or QTcF interval >460 msec.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (9):
- United States (4):
  - Dept of Obstetrics and Gynecology, Medical College of Georgia, Augusta, Georgia
  - Division of Gynecologic Oncology, University of Minnesota Medical Center, Minneapolis, Minnesota
  - Jordan Center for Gynecologic Cancer at Penn, University of Pennsylvania, Philadelphia, Pennsylvania
  - Crozer Chester medical Center, Upland, Pennsylvania
- Canada (5):
  - London Health Sciences Centre, University of Western Ontario, London, Ontario
  - Department of Oncology, Ottawa Cancer Center, Ottawa, Ontario
  - Dept of Obstetrics and Gynecology, Princess Margaret Hospital, Toronto, Ontario
  - CHUM-Hospital Notre-Dame Service de Gynecologic Oncologique, Montreal, Quebec
  - Department of Oncology, McGill University, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from United States of America and Canada from 08-Feb-2011. Terminated on 06-Jun-2011 and Study Completion was on 26-Jul-2011.
Pre-assignment Details: Six patients from five centres were screened for inclusion. All six patients were enrolled and treated
Period: Overall Study
Arm/Group | BN83495
Started | 6
Completed | 0
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Investigator's Decision | 1
Not completed — Disease Progression | 4

BASELINE CHARACTERISTICS:
Arm/Group | BN83495
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Sex/Gender, Customized [Number; unit: participants]
  Female | 6
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian / White | 3
  Asian | 1
  Black / African American | 1
  Unknown | 1
Region of Enrollment [Number; unit: participants]
  Canada | 4
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Determination of Clinical Benefit (CB), Defined as Sum of Patients Who Present Complete Response (CR), Partial Response (PR) or Stable Disease (SD) ≥12 Weeks (CB=CR+PR+SD≥12 Weeks) Using Response Evaluation Criteria in Solid Tumors (RECIST Version1.1)
Description: CR defined as: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  PR defined as: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  SD defined as: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (PD), taking as reference the smallest sum diameters while on study.
  PD defined as: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: 12 weeks
Population: The study was terminated early and due to the low number of patients enrolled, data was not collected/analysed for this endpoint
Arm/Group | BN83495
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: Up to 28 days after last dose
Population: All Screened Population
Measure: Number; unit: participants
Arm/Group | BN83495
Number analyzed (Participants) | 6
participants | 6

3. Secondary Outcome: Determination of Time to Progression (TTP) in This Patient Population
Description: Time to Progression (TTP): Time from first study treatment to first documentation of objective tumour progression.
Time Frame: After the last enrolled patient has been followed for at least 6 months or has progressed or died
Population: as for outcome 1
Arm/Group | BN83495
Number analyzed (Participants) | 0

4. Secondary Outcome: Determination of Progression Free Survival (PFS) in This Patient Population
Description: Progression Free Survival (PFS): Time from first study treatment until objective tumour progression or death from any cause.
Time Frame: After the last enrolled patient has been followed for at least 6 months or has progressed or died
Population: as for outcome 1
Arm/Group | BN83495
Number analyzed (Participants) | 0

5. Secondary Outcome: Determination of Overall Response Rate (ORR) in This Patient Population
Description: Overall Response Rate (ORR): Defined as the sum of CR and PR.
Time Frame: After the last enrolled patient has been followed for at least 6 months or has progressed or died
Population: as for outcome 1
Arm/Group | BN83495
Number analyzed (Participants) | 0

6. Secondary Outcome: Determination of Duration of Response in This Patient Population
Description: Duration of Response (DR): Time from the first documentation of objective tumour response (defined as CR or PR) to the first documentation of objective tumour progression or death on study due to any cause.
Time Frame: After the last enrolled patient has been followed for at least 6 months or has progressed or died
Population: as for outcome 1
Arm/Group | BN83495
Number analyzed (Participants) | 0

7. Secondary Outcome: Determination of Overall Survival in This Patient Population
Description: Overall Survival (OS): Defined as the time from first study treatment to death due to any cause.
Time Frame: 2 years after the last patient enrolled
Population: as for outcome 1
Arm/Group | BN83495
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 28 days after last dose
Description: Treatment emergent Adverse Events (TEAEs) that were reported by more than one patient.
Arm/Group | BN83495
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BN83495 (N=6)
Subdural hematoma (Injury, poisoning and procedural complications) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BN83495 (N=6)
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Vaginal discharge (Reproductive system and breast disorders) | 3
Fatigue (General disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2

LIMITATIONS AND CAVEATS:
Study terminated due to poor enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No